CLINICAL TRIAL: NCT01925638
Title: An Open-label Study in Healthy Male Subjects to Assess the Effect of a Strong CYP3A4 Inhibitor, Ketoconazole, on the Pharmacokinetics of Refametinib
Brief Title: Effect of Ketoconazole on the Pharmacokinetics of Refametinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14751
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Drug Interactions
Keywords: Healthy Volunteers; Refametinib; Ketoconazole; Pharmacokinetics
MeSH Terms: interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY86-9766 (Experimental): The study will be conducted in two parts and study treatments will be administered as follows: •Part A: Three subjects will be enrolled and will receive 10 mg of refametinib on Day 1. Once daily dosing of ketoconazole 400 mg will be initiated on Day 5 and will continue until Day 12 with 10 mg of refametinib administered concomitantly on Day 8 •Part B: Fifteen subjects will be enrolled and will receive refametinib doses of 10 mg, 20 mg or 30 mg on Days 1 and 8 with the same dose administered on both days. Refametinib dose for Part B will be based on safety and refametinib pharmacokinetics in Part A. Ketoconazole 400 mg will be administered once daily on Days 5 to 12. Subjects will stay in the investigational site for a total period of 15 consecutive days
  Interventions: Drug: BAY86-9766; Drug: Ketoconazole

INTERVENTIONS:
Drug: BAY86-9766
Drug: Ketoconazole

SUMMARY:
The purpose of this study is to see if there is a difference between the way your body absorbs and distributes BAY86-9766 when given alone or in combination with ketoconazole, a drug which may affect how much BAY86-9766 is absorbed, distributed or eliminated from the body

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening examination / visit
* Body mass index (BMI): 18.5 to 32 kg/m² (inclusive)
* Ability to understand and follow study-related instructions. Subject, who is a sexually active man and has not been surgically sterilized, must consent that he uses a condom during intercourse and ensures that his female partner practices adequate contraception, or he must be willing to refrain from sexual intercourse from the beginning of the trial (signing of the informed consent) until 30 days after last study drug administration

Exclusion Criteria:

* Clinically significant disease or condition
* Retinal pathology or vien occlusion
* Left Ventricular ejection Fraction(LVEF) <60% (as measured at screening) by Multiple Gated Acquisition Scan(MUGA) or echocardiogram

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cmax(maximum observed drug concentration in measured matrix after single dose administration) of BAY86-9766 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
AUC(area under the concentration vs. time curve from zero to infinity after single (first) dose) of BAY86-9766 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
t1/2(half-life associated with the terminal slope) of BAY86-9766 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 2.5 months
AUC(0-tlast)(AUC from time 0 to the last data point > LLOQ) of BAY86-9766 and Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
tmax(time to reach Cmax) of BAY86-9766 and Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
tlast(time of last observed concentration value above lower limit of quantitation) of BAY86-9766 and Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
Cmax(maximum observed drug concentration in measured matrix after single dose administration) of Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
AUC(area under the concentration vs. time curve from zero to infinity after single (first) dose) of Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
t1/2(half-life associated with the terminal slope) of Metabolites M-11 and M-17 | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
CL/F(total body clearance of drug calculated after extravascular administration) of BAY 86-9766) | Day 1: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 and 96 h post-dose; Day 8: pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States